CLINICAL TRIAL: NCT03417375
Title: Assessment of the Quality and Quantity of Bone Regeneration in the Maxillary Sinus Using Osteocel With Scaffold or Allograft Materials: A Radiographic and Histomorphometric Randomized Controlled Clinical Study.
Brief Title: Assessment of the Quality and Quantity of Bone Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmad Kutkut (Other)
Responsible Party: Sponsor-Investigator, Ahmad Kutkut, Associate Professor, Restorative Dentistry, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0102-F2L
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Bone Quality and Quantity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Osteocel Plus (Experimental): Experimental product will be placed in one sinus while the control product will be placed in the contralateral sinus. (Randomized)
  Interventions: Procedure: Bilateral Sinus Augmentation
- alloOss (Active Comparator): The control product will be placed in one sinus while the control product will be placed in the contralateral sinus. (Randomized)
  Interventions: Procedure: Bilateral Sinus Augmentation

INTERVENTIONS:
Procedure: Bilateral Sinus Augmentation — Lateral window sinus augmentation with core samples harvested from the window following 4 months of healing.

SUMMARY:
The purpose of this study is to histologically and radiographically evaluate the maxillary sinus bone volume and density, with reference to percentage of vital bone present, after four months of grafting with either Osteocel or a cortical-cancellous allograft.

1. To assess the quality and quantity of the maxillary sinus bone prior to the placement of dental implants and subsequent restorations, approximately 20 patients will be randomly assigned to receive an augmentation of the maxillary sinus region using either Osteocel or a cortical-cancellous allograft.
2. With the use of pre-operative and four months post-operative CBCT radiography, the maxillary sinus bone density will be assessed and compared between the individuals receiving Osteocel and the individuals receiving conventional cortical-cancellous allograft material.
3. Histomorphometric analysis will be used to assess, compare and contrast the quality and the quantity of the new vital bone cells generated when using these different graft materials

DETAILED DESCRIPTION:
Eligible patients will be randomly assigned into one of two treatment groups using a randomization table generated by a computer. The test group (10 sinuses) will receive Osteocel Plus and control group (10 sinuses) will receive conventional cortical-cancellous particulate allograft material. The objective of this research is to serve as a pilot study, gathering information that will guide the design of a larger subsequent study. Little is known about the distribution of bone quality changes in patients who receive Osteocel Plus graft to augment the maxillary sinus. Ten subjects per group is reasonable for a pilot study, providing an 89% probability of estimating the true mean for bone quality and implant stability to within half a standard deviation in each group. These means, along with the observed standard deviations and within-subject correlations that the investigators obtain will prove essential for designing the larger, confirmatory study that constitute the next phase of this research.

A clinical radiographic/surgical guide will be fabricated for each patient to be used for CBCT scan prior to sinus augmentation procedure. The same clinical radiographic/surgical guide will be used for CBCT scan prior to the implant placement to measure the amount of bone regeneration following four months of healing at the exact sites. One line will measure the horizontal width and the other line will measure the vertical height. The horizontal width will be measured at a vertical height of 10 mm from the sinus floor in the sinus cavity based on the conventional average length of dental implant used in implant dentistry. The difference in the measurements for all surgical sites after the grafting procedure and before the implant placement will provide a clinical assessment of the amount of bone regeneration.

Forty trephined core samples will be retrieved surgically from two areas of the grafted lateral window at the time of implant placement. One core sample will be retrieved from the anterior area, approximately 4 mm distal to the anterior tack which was used to fix the resorbable membrane, and the other one will be retrieved from the posterior area, approximately 4 mm mesial of the posterior tack which was used to fix the resorbable membrane. Histomorphometric analysis will be performed on three fields for each section using specialized software. Volume of vital bone, graft remnants, and connective tissue will be measured based on the averages of the percentages at a magnification of 63X. Data will be statistically analyzed using Statistical Package for the Social Sciences (SPSS 13.0 for Windows software) program to compare between test and control groups.

ELIGIBILITY:
Inclusion Criteria:

Must be 22 years old or older. Must have at least one edentulous posterior site requiring grafting. Must have an implant restoration to replace at least one tooth in the edentulous site.

Must be available for the follow-up examinations.

Exclusion Criteria:

Current smokers Dental infections of bone Untreated periodontal disease Pregnant patients or those who are nursing Uncontrolled diabetes (via patient reported A1C) Chemotherapy/Radiation patients Autoimmune diseases Kidney disease Liver disease

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Quality of Bone Regeneration (Number of Osteoblasts per histologic section) | 4 months post-operative of sinus augmentation.
  Core samples of bone will be evaluated histomorphometrically for number of osteoblasts present.
Quantity of Bone Regeneration (Linear measurements) | 3.5 months post-operative of sinus augmentation.
  Linear measurement of HEIGHT of bone gain
Quantity of Bone Regeneration (Linear measurements) | 3.5 months post-operative of sinus augmentation.
  Linear measurement of WIDTH of bone gain
Quantity of Bone Regeneration (Linear measurements) | 3.5 months post-operative of sinus augmentation.
  Linear measurement of DEPTH of bone gain

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky College of Dentistry, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No